CLINICAL TRIAL: NCT00429026
Title: Adaptive Randomization of Fludarabine-Melphalan Versus Fludarabine-Cyclophosphamide Conditioning Regimen in Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation Using HLA-Matched Related Donor for Metastatic Renal Cell Carcinoma
Brief Title: Conditioning Regimen in Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual, study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0364
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2009-07-13 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Renal Cell Cancer
Keywords: Kidney Cancer; Renal Cell Cancer; Stem Cell Transplant; Cyclophosphamide; Fludarabine; Melphalan; NST
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — fludarabine; Melphalan; Cyclophosphamide; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine + Cyclophosphamide with ASCT (Experimental): ASCT=Allogeneic Hematopoietic Stem Cell Transplantation
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Stem Cell Transplant
- Fludarabine + Melphalan with ASCT (Experimental): ASCT=Allogeneic Hematopoietic Stem Cell Transplantation
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 intravenous (IV) daily for 5 Days
Drug: Melphalan — 70 mg/m^2 IV Daily for 2 Days
  Arms: Fludarabine + Melphalan with ASCT
Drug: Cyclophosphamide — 60 mg/kg IV Daily for 2 Days
  Arms: Fludarabine + Cyclophosphamide with ASCT
Procedure: Stem Cell Transplant — Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation Using HLA-Matched Related Donor
  Other Names: ASCT

SUMMARY:
Primary Objectives:

1. To compare the overall survival of metastatic renal cell carcinoma (RCC) patients undergoing HLA-matched related donor nonmyeloablative allogeneic hematopoietic stem cell transplantation (NST) using fludarabine-melphalan (FM) versus fludarabine-cyclophosphamide (FC) conditioning regimen.
2. To assess both cytotoxic T lymphocyte reactivity and antibodies activity against potential tumor antigenic peptides involved in graft-versus-RCC effect.

Secondary Objectives:

1. To study the patient characteristics of metastatic RCC patients who undergo NST and those who do not undergo NST.
2. To compare the incidence of Day-100 treatment-related mortality in FM group and FC group.

DETAILED DESCRIPTION:
Registration:

When you are willing to undergo stem cell transplantation for kidney cancer, have possible related donors, and the study doctor decides you are eligible to participate, you will be enrolled in this study.

Before treatment begins, you will have a complete physical exam, including blood (about 1-2 tablespoons) and urine tests. An electrocardiogram (ECG--a test to measure the electrical function of the heart) and a heart scan will be done. A test of lung function will be done. This will involve blowing into a machine that records your lung capacity. Tissue typing will also be done by blood test on you and your possible donors to find out if you have a donor or not. Women who are able to have children must have a negative blood test in order to participate.

If you have a suitable related donor, have financial approval for the transplant procedure, and are still eligible in this study, you will go for the stem cell transplantation. A separate informed consent about the transplant procedure will be provided to you. You will need to sign and agree with the second informed consent before the start of treatment. This informed consent is only for you to be enrolled and registered in the study.

If you have no suitable related donor, no financial approval for the transplant procedure, and/or you refuse to undergo transplant for non-medical reasons, you will not have a stem cell transplant but will still remain in our study. You can receive any form of non-transplant treatment from your physician. Study researchers will only follow your progress, so that in the future, they can compare your progress with those who had the stem cell transplant.

This is an investigational study. About 480 patients will take part in this study. All patients will be enrolled at M. D. Anderson Cancer Center.

Treatment:

The two different chemotherapy regimens used in this study are fludarabine and melphalan, or fludarabine and cyclophosphamide. They act by suppressing our immune system and make space in our bone marrow so as to prepare for the new bone marrow to grow.

Before treatment starts, you will have a complete physical exam, including blood (about 1-2 tablespoons) and urine tests. An electrocardiogram (ECG-a test to measure the electrical activity of the heart) and a heart scan will be done. A test of lung function will be done. This will involve blowing into a machine that records your lung capacity. Tests will be performed to look at the status of your cancer, including chest x-ray, bone scan, CT scans, and MRI scan if needed. You will have a dental exam. Women who are able to bear children must have a negative blood pregnancy test in order to participate.

In this study, you will receive high-dose chemotherapy to prepare for the blood stem cell transplant. Two different types of chemotherapy will be used. You will be assigned to receive one of the chemotherapy treatments. As the study moves forward, the group treatment that is shown to be more effective will receive more new participants than the other one. The first chemotherapy treatment is a combination of fludarabine and melphalan. The second chemotherapy treatment is a combination of fludarabine and cyclophosphamide. The drug fludarabine will be given through a needle in your vein on Days 1-5. Depending on which treatment group you are assigned to, the drugs melphalan or cyclophosphamide will be given through a needle in your vein on Days 4 and 5, along with your scheduled dose of fludarabine. Day 6 will be a rest day; no drugs will be given. The stem cell transplant will be performed on Day 7. Bone marrow from the donor may be used instead of blood stem cells, if the collection of blood stem cells is not enough. A catheter (a tube) will be placed in a large vein in your chest to decrease the number of times you are stuck with a needle.

Blood stem cells will be collected from your family member, who has been using G-CSF to prepare for the transplant. They will need to have enough stem cells before transplantation.

The drugs tacrolimus and methotrexate will be given to ease side effects after the transplant. Tacrolimus is given by vein or by mouth for 2 to 3 months after the transplant. During the last month it is given, the dose will be decreased gradually. Methotrexate is given by vein on Days 1, 3, and 6 after the transplant. An extra dose of methotrexate will be given on Day 11, if your donor is your parent or child. Blood transfusions may be needed also.

Sometimes, the transplanted cells attack the normal cells in your body instead of the cancer cells. This is called graft-versus-host disease (GVHD). The drug methylprednisolone will be given by vein or by mouth to fight GVHD if it happens.

You must stay in the hospital for about 3 to 4 weeks. You must stay in the Houston area for about 100 days after the transplant. Blood tests (about 1-2 tablespoons) will be done every day while you are in the hospital. Chest x-rays, CT scans, and bone scans will be done once a month during the 100 days, and then every 3 months for the first year after that, so that researchers can follow your disease response.

If there are no signs of disease after 100 days, treatment will stop. You must return to the clinic for checkups every 3 months for the first year, then 3 times a year for the next 4 years, and once a year after that. If the disease is still present after 2 months, but you do not have GVHD, the anti-rejection medicine tacrolimus will be stopped within 2 weeks. Then if the disease is still present after another 6 weeks, but you do not have GVHD, you may receive an injection of donor lymphocytes by vein. This treatment may be repeated up to 3 times, with 6 weeks between each time.

If no disease is found or if GVHD occurs, treatment will stop.

This is an investigational study. About 80 participants enrolled in this study will take part in the stem cell transplant. All will be enrolled at M. D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. For registration: Willing to undergo allogeneic transplantation.
2. For registration: Age equal to or less than 65 years old.
3. For registration: Metastatic RCC with predominant conventional cell type.
4. For registration: Prior nephrectomy.
5. For registration: Stage IV RCC. If patient has prior single brain metastasis treated with complete surgical resection or stereotactic radiation therapy, no recurrence or brain edema from the end of treatment for at least 6 months has to be shown by radiological imaging.
6. For registration: Zubrod performance status < one.
7. For registration: Potential related donor for allogeneic stem cell transplantation.
8. For registration: At least one prior treatment for metastatic RCC. Radiation therapy or surgery is not counted as a treatment.
9. For registration: Signed an informed consent.
10. For transplantation: Zubrod performance status < one.
11. For transplantation: An HLA-matched (defined as 6/6 matches) related donor.
12. For transplantation: Failed at least one prior treatment for metastatic RCC. Radiation therapy or surgery is not counted as a treatment.
13. For transplantation: Adequate major organ functions (see section 4.17-4.20).
14. For transplantation: Signed an informed consent for allogeneic stem cell transplantation.

Exclusion Criteria:

1. For registration: Prior history of allogeneic stem cell transplantation.
2. For registration: Histologic feature with predominant non-conventional cell type.
3. For registration: Multiple brain metastasis.
4. For registration: Life expectancy is severely limited by concomitant illness.
5. For transplantation: Multiple brain metastasis.
6. For transplantation: Life expectancy is severely limited by concomitant illness.
7. For transplantation: Clinically significant active infections.
8. For transplantation: HIV infection.
9. For transplantation: Chronic active hepatitis
10. For transplantation: Pregnant or lactating women.
11. For transplantation: Has all three risk factors: high serum lactate dehydrogenase, low hemoglobin, high corrected serum calcium.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: January 16, 2004 through March 29, 2006. All participants recruited at U.T. M.D. Anderson Cancer Center.
Pre-assignment Details: Only 5 patients received allogeneic stem cell transplantation while 35 received standard chemotherapy. Study terminated due to low patient accrual. This population was not analyzed by treatment arm on this study.
Groups:
- Conditioning Regimen: Chemotherapy including combinations of Fludarabine, Melphalan, Cyclophosphamide
Period: Overall Study
Arm/Group | Conditioning Regimen
Started | 40
Completed | 0
Not Completed | 40
Not completed — Inevaluable for response. | 40

BASELINE CHARACTERISTICS:
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 40
Age Continuous [Median (Full Range); unit: years] | 48 (0) [30 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate
Description: Number of participants surviving at 4 years compared to total participants, to compare the overall survival of metastatic renal cell carcinoma (RCC) patients undergoing HLA-matched related donor nonmyeloablative allogeneic hematopoietic stem cell transplantation (NST) using fludarabine-melphalan (FM) versus fludarabine-cyclophosphamide (FC) conditioning regimen. Evaulation after 1, 2, 3, 6, 9, & 12 months, then every 4 months for 4 years.
Time Frame: Up to 4 years
Population: Primary outcome measure was not assessed due to early study termination, e.g. patients did not receive assigned treatment.
Arm/Group | Conditioning Regimen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years and 7 months
Arm/Group | Conditioning Regimen
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 5/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Regimen (N=40)
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5

LIMITATIONS AND CAVEATS:
Primary outcome measure was not assessed due to early study termination, e.g. patients did not receive assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No